CLINICAL TRIAL: NCT06500676
Title: An Open-Label, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of GFH375 in Patients With KRAS G12D Mutant Advanced Solid Tumors
Brief Title: A Study of GFH375 in Patients With Advanced Solid Tumors With KRAS G12D Mutations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH375X1101
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: KRAS G12D Mutations; Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GFH375 (Experimental)
  Interventions: Drug: GFH375

INTERVENTIONS:
Drug: GFH375 — GFH375 will be administered at the assigned dose level, orally, until disease progression or intolerable toxicity.

SUMMARY:
This is a multicenter, open-label, phase I/II study to explore the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of GFH375 in patients with advanced solid tumors harboring a KRAS G12D mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
2. Male or female ≥ 18 years old and ≤75 years old.
3. ECOG performance status of 0-1.
4. With a life expectancy of ≥12 weeks.
5. With histologically or cytologically confirmed advanced or metastatic solid tumors harboring KRAS G12D mutation.
6. Have at least one measurable lesion according to RECIST1.1, and the phase Ia allows no measurable lesion.
7. Adequate laboratory parameters during the screening period.

Exclusion Criteria:

1. Active brain metastases.
2. Prior treatment with a KRAS G12D inhibitor.
3. Palliative radiotherapy was completed within 14 days before the first dose.
4. Have poorly controlled or severe cardiovascular disease.
5. Subjects with active hepatitis B or active hepatitis C.
6. Known allergy to the study drug or its components.
7. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ia:The incidence and severity of AEs and SAEs | 24 months
  The incidence and severity of AEs and SAEs
Phase Ia:The incidence of DLT events | 21 days
  The incidence of DLT events
Phase Ib:The incidence and severity of AEs and SAEs | 24 months
  The incidence and severity of AEs and SAEs
Phase II:Overall response rate (ORR) | 24 months
  For NSCLC cohort： Assessed by BICR according to RECIST 1.1；For other cohorts： Assessed by investigators according to RECIST 1.1；

SECONDARY OUTCOMES:
Plasma concentrations | up to 21 days
  Plasma concentrations and PK parameters of GFH375
Efficacy endpoints | 24 months
  Duration of response (DoR)
Efficacy endpoints | 24 months
  Disease control rate (DCR)
Efficacy endpoints | 24 months
  Progression free survival (PFS)
Efficacy endpoints | 24 months
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital; Aiping Zhou, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (20):
- China (20):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Chest Hospital, Shanhai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing, Tianjing
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No